CLINICAL TRIAL: NCT07398040
Title: Clinical Impact of an Anti-Inflammatory Diet in Anxiety and Depression Detected by an AI-Based Screening Model
Brief Title: Clinical Impact of an Anti-Inflammatory Diet in Anxiety and Depression With AI
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Zaragoza (Other)
Responsible Party: Principal Investigator, María Isabel Iguacel Azorín, Dr, Universidad de Zaragoza
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Anti-inf-AI
Record Dates: First submitted 2026-01-13; First posted 2026-02-09 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Depression - Major Depressive Disorder; Anxiety
Keywords: Depression; Anxiety; Anti-inflammatory diet; Artificial Intelligence
MeSH Terms: conditions — Anxiety Disorders; Depression

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Anti-inflammatory diet (Experimental)
  Interventions: Other: Anti-inflammatory diet
- Control (Active Comparator)
  Interventions: Other: Control

INTERVENTIONS:
Other: Anti-inflammatory diet — We will use an anti-inflammatory diet to assess its impact on physical, mental and cognitive health
  Arms: Anti-inflammatory diet
Other: Control — No intervention
  Arms: Control

SUMMARY:
The goal of this clinical trial is to evaluate the effectiveness of an anti-inflammatory dietary intervention on physical health, mental health, and cognitive functioning in individuals with clinically diagnosed anxiety and/or depression, and to assess the agreement between artificial intelligence-based analysis of verbal and non-verbal language patterns and standard psychometric assessment tools.

The study will include adult participants (≥18 years) with a clinical diagnosis of anxiety and/or depressive disorder, irrespective of sex or gender.

The main questions it aims to answer are:

Does a 4-month anti-inflammatory dietary intervention improve mental health outcomes (anxiety and depressive symptoms) compared to a control condition in individuals with anxiety and/or depression?

Does the intervention lead to improvements in physical health and cognitive functioning relative to the control group?

Are verbal and non-verbal language patterns analyzed using artificial intelligence coherent with the results obtained from validated anxiety and depression questionnaires at baseline?

Do changes in AI-derived language markers parallel changes in clinical and self-reported outcomes following the dietary intervention?

Primary outcomes / hypotheses:

Does the anti-inflammatory dietary intervention produce greater reductions in anxiety and depressive symptom severity compared to the control group after 4 months?

Does the intervention result in significant improvements in physical health and cognitive performance compared to the control group?

Researchers will compare the anti-inflammatory diet intervention group with the control group (usual diet or standard dietary advice) to determine whether the intervention leads to superior improvements in mental, physical, and cognitive health outcomes.

Participants will:

Complete baseline assessments including validated questionnaires on anxiety, depression, physical health, cognitive functioning, and quality of life.

Undergo structured interviews at baseline during which verbal and non-verbal language data will be recorded and analyzed using artificial intelligence-based models.

Be allocated to either the anti-inflammatory dietary intervention group or the control group.

Follow their assigned dietary condition for 4 months.

Complete post-intervention assessments identical to baseline, including psychometric questionnaires and cognitive and physical health evaluations.

ELIGIBILITY:
- Inclusion Criteria: Age 18 years or older.

Presence of mild, moderate, or severe symptoms of anxiety, depression, or stress, as measured by the DASS-42 questionnaire.

Absence of medical contraindications to following a personalized diet.

Absence of cognitive impairment.

Proficiency in the Spanish language (ability to speak and understand fluently).

Availability over a 4-month period to attend scheduled assessments and intervention sessions.

Low or moderate adherence to the Mediterranean diet, as assessed by the Mediterranean Diet Adherence Questionnaire (score ≤ 9 out of 14).

Residence in the city of Zaragoza for the entire duration of the study.

Signed informed consent after receiving detailed information about the study.

- Exclusion Criteria: DASS-42 scores compatible with either extremely severe symptomatology (requiring urgent clinical care) or with normal-range results.

Presence of organic pathologies that prevent adherence to the dietary intervention or that significantly interfere with the conduct of the study.

Inability to attend the scheduled in-person sessions.

Diagnosis or suspicion of a clinically unstable systemic medical disorder, or a physical illness currently causing severe physical and/or mental distress (e.g., an active flare of inflammatory bowel disease).

Pregnancy.

Current participation in another specific intervention focused on diet or exercise.

Diagnosis of severe psychiatric disorders, such as bipolar disorder type I or II, or a personality disorder as the primary clinical diagnosis.

Current substance use disorder.

Medical diagnosis that could explain or mask potential psychopathology, such as hormonal alterations (e.g., uncontrolled thyroid dysfunction).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2026-01-16 (Estimated); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Anxiety level (Depression, Anxiety, Stress Scale; DASS-42) | From enrollment to the end of treatment at 16 weeks
Depression level (Depression, Anxiety, Stress Scale; DASS-42) | From enrollment to the end of treatment at 16 weeks
SF-36 | From enrollment to the end of treatment at 16 weeks
GLUCEMIC PROFILE | From enrollment to the end of treatment at 16 weeks
INFLAMMATORY PROFILE | From enrollment to the end of treatment at 16 weeks

SECONDARY OUTCOMES:
Gastrointestinal symptoms (Gastrointestinal Symptom Rating Scale) | From enrollment to the end of treatment at 16 weeks
Physical activity (International Physical Activity Questionnaire) | From enrollment to the end of treatment at 16 weeks
  We evaluate intense, moderate and soft physical activity through IPAQ questionnaire
Sleep quality (Pittsburg Sleep Quality Index) | From enrollment to the end of treatment at 16 weeks
Food Frequency Questionnaire | From enrollment to the end of treatment at 16 weeks
Adherence to Mediterranean diet (MEDAS Scale) | From enrollment to the end of treatment at 16 weeks
  We evaluate the adherence to the mediterranean diet through MEDAS scale
BMI | From enrollment to the end of treatment at 16 weeks
Weight | From enrollment to the end of treatment at 16 weeks
CD-RISK | From enrollment to the end of treatment at 16 weeks
LIPID PROFILE | From enrollment to the end of treatment at 16 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Universidad of Zaragoza, Zaragoza, Zaragoza, Spain

IPD SHARING:
Plan to Share IPD: No